CLINICAL TRIAL: NCT01759511
Title: A Phase 2, Long-Term Safety Study of GS-6624 in Adult Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Long-Term Safety Study of GS-6624 in Adults With Idiopathic Pulmonary Fibrosis (IPF)
Acronym: ATLAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Study was terminated due to lack of efficacy.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-322-0206
Record Dates: First submitted 2012-11-15; First posted 2013-01-03 (Estimated); Results first posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic; Pulmonary; Fibrosis; IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Fibrosis | interventions — simtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Simtuzumab (Experimental): Participants will receive simtuzumab.
  Interventions: Drug: Simtuzumab

INTERVENTIONS:
Drug: Simtuzumab — 200 mg/mL administered intravenously biweekly (per original protocol) or 125 mg/mL self-administered subcutaneously every 7 ± 2 days (per protocol amendment 1)
  Other Names: GS-6624

SUMMARY:
The primary objective of this study is to evaluate the long term safety and tolerability of simtuzumab (GS-6624) in participants with idiopathic pulmonary fibrosis (IPF) who had previously participated in Gilead clinical trial AB0024-201.

ELIGIBILITY:
Key Inclusion Criteria:

* Previous participation in Phase 1 Gilead clinical trial
* Diagnosis of idiopathic pulmonary fibrosis
* Females of childbearing potential and non-vasectomized males must agree to use highly effective methods of contraception
* Females must discontinue nursing
* Comply with study requirements
* Have adequate organ function

Key Exclusion Criteria:

* History or evidence of clinically significant disorder, condition or disease that would pose a risk or interfere with the study
* Pregnant or lactating
* Clinically significant heart, hepatic or renal disease
* History of cancer within 5 years of screening
* Infection that is not controlled despite antibiotics or other treatment
* History of bleeding diathesis within the last 6 months of Day 1
* Known history of human immunodeficiency virus, hepatitis B or C
* Concern's for subjects compliance
* Other conditions that might put the subject at high risk for treatment complications or reduce the chance to obtain data required
* Placed on a lung transplant list
* Previous participation in an idiopathic pulmonary fibrosis clinical trial other than for simtuzumab

Note: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-10-18 (Actual); Primary Completion 2016-02-19 (Actual); Study Completion 2016-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (6):
- United States (6):
  - Arizona Pulmonary Specialists, Ltd., Scottsdale, Arizona
  - University of California, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 6 study sites in the United States. The first participant was screened on 18 October 2012. The last study visit occurred on 19 February 2016.
Pre-assignment Details: 37 participants were screened.
Period: Overall Study
Arm/Group | Simtuzumab
Started | 34
Completed | 0
Not Completed | 34
Not completed — Adverse Event | 4
Not completed — Death | 2
Not completed — Lack of Efficacy | 2
Not completed — Physician Decision | 1
Not completed — Progressive Disease | 5
Not completed — Protocol-Specified Criteria for Withdraw | 4
Not completed — Study Terminated by Sponsor | 13
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received at least 1 dose of study drug
Arm/Group | Simtuzumab
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (7.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 34
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 33
Forced vital capacity (FVC) Percent Predicted [Mean (Standard Deviation); unit: FVC % predicted] | 69.9 (14.18)
FVC % Predicted Category [Count of Participants; unit: Participants]
  Mild | 12
  Moderate | 16
  Severe | 6
Forced expirator volume in the first second of expiration (FEV1)/FVC Ratio [Mean (Standard Deviation); unit: liter] | 0.8 (0.23)
Hemoglobin-Corrected Carbon dioxide diffusing capacity (DLCO) Predicted [Mean (Standard Deviation); unit: DLCO % predicted] | 12.2 (4.22)

OUTCOME MEASURES:

1. Primary Outcome: Overall Safety Profile of Simtuzumab
Description: The overall safety of simtuzumab was assessed as the percentage of participants experiencing adverse events (AEs; Serious AEs, Grade 3 or 4 AEs, AEs related to simtuzumab, and AEs leading to discontinuation of simtuzumab), treatment-emergent chemistry and hematology abnormality.
Time Frame: 30 days post last study treatment (up to 165 weeks)
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Simtuzumab
Number analyzed (Participants) | 34
percentage of participants
  Adverse Events (AEs) | 97.1
  Grade 3 or 4 AEs | 47.1
  Serious Adverse Events | 35.3
  SAEs Related to simtuzumab | 5.9
  AEs leading to discontinuation of simtuzumab | 29.4

2. Secondary Outcome: Relative Change From Baseline in FVC % Predicted at Weeks 72 and 144
Description: * FVC was a pulmonary function test, and was defined as the volume of air that can forcibly be blown out after taking a full breath.
  * Least square means were from mixed model for repeated measures (MMRM) model including baseline FVC % predicted and visit including all data up to Week 144.
Time Frame: Weeks 72 and 144
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in FVC % predicted
Arm/Group | Simtuzumab
Number analyzed (Participants) | 34
percent change in FVC % predicted
  Week 72: number analyzed (Participants) | 19
  Week 72 | -8.05 (1.829)
  Week 144: number analyzed (Participants) | 13
  Week 144 | -12.04 (2.086)

3. Secondary Outcome: Relative Change From Baseline in DLCO % Predicted at Weeks 72 and 144
Description: * DLCO was a measurement to determine the extent to which oxygen passes from the air sacs of the lungs into the blood.
  * Least square means were from MMRM model including baseline DLCO % predicted and visit including all data up to Week 144.
Time Frame: Weeks 72 and 144
Population: Participants in Safety Analysis Set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in DLCO % predicted
Arm/Group | Simtuzumab
Number analyzed (Participants) | 34
percent change in DLCO % predicted
  Week 72: number analyzed (Participants) | 19
  Week 72 | -7.41 (3.062)
  Week 144: number analyzed (Participants) | 13
  Week 144 | -22.80 (3.475)

4. Secondary Outcome: All-cause Mortality
Description: All-cause mortality was assessed as a number of participants who died from any cause.
Time Frame: Up to 165 weeks
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Simtuzumab
Number analyzed (Participants) | 34
Participants | 3

5. Secondary Outcome: Relative Change From Baseline in Serum Lysyl Oxidase-like 2 (sLOXL2) Levels at Weeks 72 and 120
Time Frame: Weeks 72 and 120
Population: Participants in the Safety Analysis set with available data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: percent change in sLOXL2
Arm/Group | Simtuzumab
Number analyzed (Participants) | 34
percent change in sLOXL2
  Week 72: number analyzed (Participants) | 19
  Week 72 | 5.93 (5.937)
  Week 120: number analyzed (Participants) | 16
  Week 120 | -0.69 (6.032)

ADVERSE EVENTS:
Time Frame: 30 days post last study treatment (up to 165 weeks)
Description: Safety Analysis Set
Arm/Group | Simtuzumab
All-Cause Mortality (participants affected / at risk) | 3/34
Serious Adverse Events (participants affected / at risk) | 12/34
Other Adverse Events (participants affected / at risk) | 33/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Simtuzumab (N=34)
Leukocytosis (Blood and lymphatic system disorders) | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Aortic stenosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Simtuzumab (N=34)
Anaemia (Blood and lymphatic system disorders) | 4
Tachycardia (Cardiac disorders) | 2
Cataract (Eye disorders) | 2
Dry eye (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 5
Flatulence (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Chest discomfort (General disorders) | 2
Chest pain (General disorders) | 2
Chills (General disorders) | 2
Fatigue (General disorders) | 10
Infusion site extravasation (General disorders) | 2
Injection site bruising (General disorders) | 2
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 8
Pyrexia (General disorders) | 3
Bronchitis (Infections and infestations) | 7
Gastroenteritis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Nail infection (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 3
Fall (Injury, poisoning and procedural complications) | 2
Laceration (Injury, poisoning and procedural complications) | 2
Procedural pain (Injury, poisoning and procedural complications) | 4
Blood pressure increased (Investigations) | 2
Gamma-glutamyltransferase increased (Investigations) | 2
Occult blood positive (Investigations) | 2
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 3
Mental status changes (Psychiatric disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 18
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years